CLINICAL TRIAL: NCT04821011
Title: Assessment of Autonomic Regulation During the Listening of Mother Heart Beat in Newborns
Acronym: Cardio_Sound
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN462021/CHUSTE
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-03

CONDITIONS: Premature Birth
Keywords: Premature; Maternal heart beat; Newborn; Heart rate Variability; Autonomous nervous system
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Newborn birth between 28 and 40 Weeks of Gestational Age (wGA): Newborn birth between 28 and 40 Weeks of Gestational Age (wGA) will be included. The mother's newborn will be have a record of her heartbeats.
  The newborn will be have an acoustic listening of their mother's heartbeat and a record of their own heartbeats.
  Interventions: Device: electronic stethoscope; Device: acoustic listening of mother's heartbeats; Device: Recording of the newborn's heart rate

INTERVENTIONS:
Device: electronic stethoscope — Record of maternal heart sounds (heartbeats) with an electronic stethoscope during 10 minutes.
  Other Names: Littmann® Electronic 3200
Device: acoustic listening of mother's heartbeats — Each newborn included will have 20 minutes of an acoustic listening of their mother heartbeats previously recorded.
Device: Recording of the newborn's heart rate — Recording of the newborn's heart rate: one hour before the acoustic listening, during the acoustic listening and one hour after the acoustic listening .
  The variations of the autonomic nervous system will be analyzed.
  An coupled Heart rate variability recording (ECG signal obtained from a Philips® IntelliVue MX700 monitor) and NIPΣ index of comfort (MDMS® NIPΣ monitor) will be used.
  Other Names: Philips® IntelliVue MX700 monitor; MDMS® NIPΣ monitor

SUMMARY:
Prematurity birth lead to an early breaking link with the in utero environment. A special attention is brought in the neonatal intensive care units to reduce noise and lighting surrounding aiming to protect the newborn.

During the uterine life fetus benefits previously of several auditory stimulations by the maternal voice, the mother's heartbeat. After birth the auditory environment is dramatically modified.

Aim of this study is to submit to the newborn an audio recording of his mother's heart beat to analyze the comfort, stress and autonomic response. Heart rate variability (HRV) analysis is a non-invasive tool able to consider autonomic nervous system activity. Previous studies have shown that pleasant feelings are associated with an increase of high frequencies variations index (HFnu index) reflecting a prevalence of parasympathetic activity in the sympathetic-parasympathetic balance. This one can be simply assess by a monitor named NIPΣ and can provide a comfort index by quantifying the parasympathetic tone.

DETAILED DESCRIPTION:
The study will imply 40 preterm and term newborns hospitalized in neonatal intensive care units of the University Hospital of Saint-Etienne (France).

ELIGIBILITY:
Inclusion Criteria:

* Neonates between 28 and 40 Weeks of Gestational Age (wGA)
* Hospitalized in the neonatal intensive care units of the university hospital of Saint-Etienne (France)

Exclusion Criteria:

* Respiratory or hemodynamic instability
* Uncontrolled sepsis
* Sedation on going
* Treatment known to modify the sympathetic or parasympathetic activity of the autonomic nervous system
* Congenital disease
* Congenital ear pathology

Ages: 4 Days to 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborn birth between 28 and 40 Weeks of Gestational Age (wGA) will be included.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2021-06-27 (Actual); Study Completion 2021-06-27 (Actual)

PRIMARY OUTCOMES:
NIPΣ index | During the acoustic listening
  Analyze variations of the activity of the autonomic nervous system (R-R cardiac interval)
  NIPΣ index (from 0 to 100) obtained from an MDoloris® monitor.
  The base line is measured one hour before

SECONDARY OUTCOMES:
HFnu (normalized high frequency) index. | During the acoustic listening
  Measured by analyze of record's of newborn heart rate.
  The base line is measured one hour before
HFnu (normalized high frequency) index. | One hour after the acoustic listening
  Measured by analyze of record's of newborn heart rate.
Standard deviation of all NN intervals (SDNN) | During the acoustic listening
  Measured by analyze of record's of newborn heart rate
Standard deviation of all NN intervals (SDNN) | One hour after the acoustic listening
  Measured by analyze of record's of newborn heart rate
Proportion of NN50 divided by the total number of NN intervals (pNN50) | During the acoustic listening
  Measured by analyze of record's of newborn heart rate
Proportion of NN50 divided by the total number of NN intervals (pNN50) | One hour after the acoustic listening
  Measured by analyze of record's of newborn heart rate
Root mean square of the successive differences (RMSSD).of RR interval | One hour after the acoustic listening
  Measured by analyze of record's of newborn heart rate.
Root mean square of the successive differences (RMSSD).of RR interval | During the acoustic listening
  Measured by analyze of record's of newborn heart rate.
Total power spectrum (Ptot) | During the acoustic listening
  Measured by analyze of record's of newborn heart rate.
Total power spectrum (Ptot) | One hour after the acoustic listening
  Measured by analyze of record's of newborn heart rate.
Low Frequency (LF) | During the acoustic listening
  Measured by analyze of record's of newborn heart rate.
Low Frequency (LF) | One hour the acoustic listening
  Measured by analyze of record's of newborn heart rate.
High Frequency (HF) | During the acoustic listening
  Measured by analyze of record's of newborn heart rate.
High Frequency (HF) | One hour after the acoustic listening
  Measured by analyze of record's of newborn heart rate.
Very Low Frequency (VLF) | During the acoustic listening
  Measured by analyze of record's of newborn heart rate.
Very Low Frequency (VLF) | One hour after the acoustic listening
  Measured by analyze of record's of newborn heart rate.
Ratio Low Frequency (LF) / High Frequency (HF) | During the acoustic listening
  Measured by analyze of record's of newborn heart rate.
Ratio Low Frequency (LF) / High Frequency (HF) | One hour after the acoustic listening
  Measured by analyze of record's of newborn heart rate.
Heart rate (bpm) | During the acoustic listening
  Measured by analyze of record's of newborn heart rate.
Oxygen saturation (%) | During the acoustic listening
  Measured by analyze of record's of newborn heart rate.
NIPΣ index | One hour after the acoustic listening
  Analyze variations of the activity of the autonomic nervous system (R-R cardiac interval)
  NIPΣ index (from 0 to 100) obtained from an MDoloris® monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Hugues PATURAL, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No